CLINICAL TRIAL: NCT06962423
Title: A Study on Artificial Intelligence-based Automated Biomedical Research
Brief Title: AI-driven Automated Biomedical Research
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tsinghua University (Other)
Responsible Party: Principal Investigator, Tien Yin Wong, Vice-Provost and Senior Vice-Chancellor, Tsinghua Medicine, Tsinghua University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: THU01-20250025
Record Dates: First submitted 2025-04-15; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Biomedical Research; Artificial Intelligence (AI)
MeSH Terms: interventions — Intelligent Systems

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants will complete the research task without our AI system.
- Intervention group (Experimental): Participants will complete the research task with AI system developed by our team.
  Interventions: Other: AI system

INTERVENTIONS:
Other: AI system — Participants will complete the research task with the AI system developed by out team to perform automated biomedical research.
  Arms: Intervention group

SUMMARY:
This study will evaluate the effects of the AI system developed by our team on biomedical research.

DETAILED DESCRIPTION:
It i a randomized-controlled study. Participants will be randomly assigned to the Intervention Group using our AI system and the Control Group. Both groups will perform the same biomedical research tasks and submit reports. At the end of the study, the research performance of the two groups will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥ 18 years old;
* (2) Agree to sign consent form and invest time in this study;
* (3) Able to understand and complete research tasks.

Exclusion Criteria:

* (1) Currently participating in other projects that may interfere with this research and unable to ensure participation time;
* (2) Have a history of major diseases or poor physical condition in the past three months that may affect research participation;
* (3) Unwilling or unable to understand and complete the research tasks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Research quality evaluation scale | Through study completion, an average of 1 week
  Independent senior experts will evaluate the research reports from the Intervention Group and the Control Group using a standardized 100-point Research Quality Evaluation Scale. A higher score indicates better research quality.

SECONDARY OUTCOMES:
Model performance | Through study completion, an average of 1 week
  The diagnostic accuracy, sensitivity, specificity, and area under the receiver-operating characteristic curve (AUC-ROC) will be reported to compare the performance of models generated by the Intervention Group and the Control Group.
Research time cost | Through study completion, an average of 1 week
  The time spent by the Intervention Group and the Control Group to complete tasks will be compared.
User evaluation | Through study completion, an average of 1 week
  User evaluation on the study will be assessed by Likert Scales.
Model resource consumption | Through study completion, an average of 1 week
  GPU usage rate and time and model size will be tracked and compared to evaluate the computational resource consumption of the Intervention Group and Control Group.

CONTACTS AND LOCATIONS:
Overall Officials: Tien Yin Wong, Principal Investigator — Tsinghua University
Locations (1):
- Tsinghua University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No